CLINICAL TRIAL: NCT01102205
Title: Evaluation of Oxidative Stress and Effect of Levothyroxine Treatment on Oxidative Stress in Hashimoto Disease
Status: Completed | Type: Observational
Sponsor: Vakif Gureba Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Ali Cikrikcioglu, Vakif Gureba TRH, Vakif Gureba Training and Research Hospital
Other Study IDs: tastoshashi
Record Dates: First submitted 2010-04-09; First posted 2010-04-13 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Hashimoto Disease
MeSH Terms: conditions — Hashimoto Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — after overnight fasting state,venous blood will be taken to obtain serum.speciemens stored -70 cantigrade celcius untillanalysing.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- healthy
- euthyroid hashimoto
- hypothyroid hashimoto

SUMMARY:
Oxidative stress leads to or accompanies with numerous disease. Oxidative balance in subclinical hypothyroid or euthyroid state in Hashimoto disease are not known. Effect of levothyroxine therapy on oxidative balance are also not known in hashimoto disease.

DETAILED DESCRIPTION:
oxidative stress markers will be measured initially(TAS,TOS,OSI,PARAOXONASE,ARYLESTERASA,PON1 PHENOTYPİNG,LİPİDPEROXİD).After 3 months therapy with levothyroxine measurements will be repeated except PON1 phenotyping.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years

Exclusion Criteria:

* inability to give a written consent
* other conditions and drug usage affect oxidative stress

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult with Hashimoto disease in euthyroid or subclinical hypothyroid state and healthy control.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2010-04; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Poxidative stress markers | After levotren therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet ali Cikrikcioglu, MD, Study Chair — vakif gureba TRH,fatih,istanbul,turkey.specialist in internal medicine
Locations (1):
- Vakif Gureba Training and Research Hospital, Istanbul, Turkey (Türkiye)